CLINICAL TRIAL: NCT02082743
Title: Intervention Program for Vision Care in Lower Grade Schoolchildren
Brief Title: Vision Care Intervention for Lower Grade School Children in Taiwan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Ministry of Health and Welfare, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: C1020515; HPA-MHW-C1020515 (Other Grant/Funding Number: Health Promotion Administration, Ministry of Health and Welfare, Taiwan)
Record Dates: First submitted 2014-02-23; First posted 2014-03-10 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-07

CONDITIONS: Myopia; Outdoor Activity; Policy of Recess Outside Classroom
Keywords: Myopia; Outdoor activity; Recess outside classroom
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Outdoor activity (Experimental): Outdoor activity in recess time
  Interventions: Behavioral: Outdoor activity in recess time
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Outdoor activity in recess time — Outdoor activity in recess time
  Arms: Outdoor activity

SUMMARY:
The purpose of this study is making use of school policy- recess outside classroom (ROC7-11) for increasing the time spent outdoor during recess and encouraging children spent time outdoor up to 11 hours in each week to investigate the vision change, myopia onset and progression in these schoolchildren.

ELIGIBILITY:
Inclusion Criteria:

All the students in Grade 1

Exclusion Criteria:

No

Ages: 6 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1020 (Actual)
Dates: Start 2013-10; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Cycloplegic refraction | 1 year

SECONDARY OUTCOMES:
Axial length | 1 year

OTHER OUTCOMES:
data from light meter recorder | 1 week
questionnaire | 1 week
  Children and their parents report how many hours per week in near work (such as reading, computer game, learning and practicing violin or piano) and outdoor activities

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthamology, Kaohsiung Chang Gung Memorial Hospital and Chang Gung university College of Medicine, Kaohsiung City, Taiwan